CLINICAL TRIAL: NCT01038804
Title: A Phase II, Multicenter, Open-Label, Randomized Study of YM155 Plus Docetaxel as First-Line Treatment in Subjects With HER2 Negative Metastatic Breast Cancer
Brief Title: A Study of YM155 Plus Docetaxel as First-Line Treatment in Subjects With HER2 Negative Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 155-CL-036; 2009-012439-14 (EudraCT Number)
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Metastatic; HER2 Negative; YM155
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — sepantronium; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A. YM155 plus docetaxel (Experimental)
  Interventions: Drug: YM155; Drug: Docetaxel
- B. docetaxel alone (Active Comparator)
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: YM155 — intravenous infusion
  Arms: A. YM155 plus docetaxel
Drug: Docetaxel — intravenous infusion
  Other Names: Taxotere

SUMMARY:
The purpose of this study is to evaluate survival, response rate, safety and tolerability of YM155 given in combination with docetaxel as first-line treatment in subjects with human epidermal growth factor 2 non-overexpressing (HER2 negative) metastatic breast cancer.

DETAILED DESCRIPTION:
This is an outpatient study. All subjects enrolled in this study will receive a combined regimen of YM155 and docetaxel or docetaxel alone given during 21 day cycles. Each subject will be assessed at the end of each cycle to determine if the subject can continue to the next cycle. Each subject assigned to receive YM155 in combination with docetaxel will be eligible to continue receiving the combination regimen in this study until one of the discontinuation criteria is met.

If a subject discontinues treatment with at least stable disease (SD) that subject will complete follow-up visits every 12 weeks for 2 years or until initiating another systemic anti-breast cancer treatment, exhibiting progressive disease (PD), or death.

Each subject will be contacted by the study site every 12 weeks for survival following the End of Treatment Visit. The contacts will continue until death or for no more than 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically-proven adenocarcinoma of the breast that is HER2 negative. Subjects with hormone receptor positive or negative status are eligible. Additionally, subjects with triple negative status (meaning estrogen receptor negative, progesterone receptor negative and HER2 negative) are eligible
* No prior chemotherapy regimen for metastatic breast cancer
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1 at the Baseline Visit
* The subject's life expectancy is estimated to be > 12 weeks at the Baseline Visit
* The subject must be non-pregnant and non-lactating. All sexually active subjects of childbearing potential must agree to use an adequate method of contraception throughout the study period

Exclusion Criteria:

* Hypersensitivity to docetaxel or polysorbate 80
* Neuropathy ≥ Grade 2 at the Baseline Visit
* Known brain or leptomeningeal metastasis as assessed through medical history review and physical examination
* The subject has known Human Immunodeficiency Virus (HIV), Hepatitis B surface Antigen or hepatitis C antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2009-12; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | At the time of progression or death or at 2 year follow up

SECONDARY OUTCOMES:
Objective response rate (proportion of subjects with complete response or partial response) | At the time of progression or death or at 2 year follow up
Overall survival | At the time of death or at 2 year follow up
Duration of response | At the time of progression or at 2 year follow up
Clinical benefit rate | At the time of progression or death or at 2 year follow up
Time to response | At the time of response or at 2 year follow up
Safety assessed by recording of adverse events, physical examinations, vital signs, laboratory assessments and electrocardiograms (ECGs) | Up to 30 days after last subject discontinues treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Medical Director, Study Director — Astellas Pharma Global Development; United Kingdom Principal Investigator, Principal Investigator — Royal Bournemouth Hospital; Poland Principal Investigator, Principal Investigator — Centrum Onkologii-Instytut im.; Ireland Principal Investigator, Principal Investigator — St Vincent's University Hospital, Ireland; Germany Principal Investigator, Principal Investigator — Luisenkrankenhaus Duesseldorf; Czech Republic Principal Investigator, Principal Investigator — Thomayer Faculty Hosptial L.G.; Belgium Principal Investigator, Principal Investigator — Institut Jules Bordet - Medical Oncology and Translational Research
Locations (30):
- United States (7):
  - Kenmar Research Institute, Los Angeles, California
  - Bay Area Cancer Research Group, Pleasant Hill, California
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Karmanos Cancer Institute, Detroit, Michigan
  - Montana Cancer Institute Foundation c/o Montana Cancer Specialists, Missoula, Montana
  - Carolina Oncology Specialists, PA, Hickory, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
- Belgium (3):
  - Institut Jules Bordet - Medical Oncology and Translational Research, Brussels
  - Grand Hopital de Charleroi - Site Notre Dame, Charleroi
  - Sint-Augustinus GZA Ziekenhuizen, Wilrijk
- Czechia (2):
  - FN Kralovske Vinohrady, Prague
  - Faculty Hospital Na Bulovce, Prague
- Germany (4):
  - Hämatologisch-onkologische Praxis, Augsburg
  - Frauenklinik des Universitätsklinikums Erlangen, Erlangen
  - Universitatsklinikum Schleswig, Kiel
  - Klinikum Mutterhaus der Borromaeerinnen, Trier
- Ireland (3):
  - St. Vincent's University Hospital, Dublin
  - St. James Hospital, Dublin
  - Department of Medical Oncology, Dublin
- Poland (2):
  - Centrum Onkologii-Instytut im., Warsaw
  - Wojewodzki Szpital, Wroclaw
- Russia (8):
  - State Therapeutic and Prophylactic Institution Chelyabinsk Regional Clinical Oncology Dispensary, Chelyabinsk
  - State Healthcare institution "Kursk Regional Oncology Dispensary" of Kursk Region Healthcare committee GUZ "KOOD", Kursk
  - Institution of Russian Academy of Medical Sciences Russian Oncology Research Centre, Moscow
  - Pyatigorsk Oncology Dispensary, Pyatigorsk
  - Scientific-Research Institute of Oncology named after Petrov, Saint Petersburg
  - Saint-Petersburg State Medical University named after Pavlov, Saint Petersburg
  - State Healthcare Institution "Samara Regional Clinical Oncology Dispensary", Samara
  - Tula Regional Dispensary, Tula
- Nottingham University Hospital, Nottingham, United Kingdom